CLINICAL TRIAL: NCT02627976
Title: The Effect of Wearing a Compression Vest on Patient Reported Pain, Quality of Life and Degree of Breast Edema.
Brief Title: Breast Edema Compression Vest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Thuasne (Industry)
Responsible Party: Principal Investigator, M.L. Gregorowitsch, MD, PhD student, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL53275.041.15
Record Dates: First submitted 2015-12-04; First posted 2015-12-11 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Edema; Lymphedema; Breast Neoplasm; Breast Cancer
MeSH Terms: conditions — Edema; Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- breast edema vest (Active Comparator)
  Interventions: Device: Compression vest, Thuasne

INTERVENTIONS:
Device: Compression vest, Thuasne — Wearing a compression 4 days/weel with a minumum of 6 hours per day

SUMMARY:
A common complication of breast conserving therapy is breast edema, which may lead to chronic pain, but also reduced quality of life (QoL) and poor cosmetic outcome. When pain is present most patients are currently treated with physical therapy, but evidence of its effectiveness is still low and a gold standard does not yet exist. A downside of physical therapy is that patients have to undergo the therapy regularly and treatment might even has to continue for years after symptoms and treatment started. Another treatment option is a compression vest with the potential, apart from reducing symptoms, to improve self-efficacy in patients because they decide when to wear it without the need to visit therapists. However effectiveness of the compression vest has not yet been objectified in studies.

The aim of this pilot study is to study if there is an effect on pain, QoL and the amount of breast edema of wearing a compression vest, in order to determine whether a large randomized study is feasible.

DETAILED DESCRIPTION:
In this pilot study, a maximum of 40 patients with symptomatic breast edema after surgery and/or radiotherapy for breast cancer are offered treatment with a compression vest. These patients will be followed for 6 months. Recruitment will continue until 20 active vest users are participating.

Primary endpoint is the course of patient reported pain over a 6 month period. Secondary endpoints are the course of degree of breast edema and quality of life over a 6 month period.

Patients who are wearing the vest may experience relief of breast edema related symptoms. In terms of burden, they might experience a tight feeling on the skin while wearing the vest, which could also be the case when treated with compression therapy and taping by a physical therapist. This tight feeling can be overcome by changing the vest to a larger size. All patients will fill out questionnaires upon inclusion, at 2 weeks, and 1, 3 and 6 months. This will take approximately 10-15 minutes per follow-up moment. Patients will have to visit the hospital at baseline and 1, 3 and 6 months after they started wearing the vest (i.e. 25 minute consult with physical examination, photo documentation of the breast and short basic follow-up questions), and it is expected that additional measurements for fitting a new compression vest will need to be taken 2-5 times during participation in the study. Those fitting measurements will be performed at a location as desired by the patient (e.g. UMC Utrecht or at patients' home).

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 18 years and older.
* Patient treated with surgery and/or radiotherapy for breast cancer, with symptomatic breast edema (e.g. pain).
* Visual Analog Scale (VAS) pain score of 3 or more.

Exclusion Criteria:

* Inability to understand the Dutch language.
* Indicated to undergo radiation treatment of the breast/chestwall within the next 6 months.
* Cardiac complaints.
* Pacemaker.
* Port-a-cath.
* Thrombosis of the arm.
* Pulmonary embolism.
* Pulmonary disease.
* Pregnancy.
* Non-breast cancer related lymph edema.
* Clinical depression or anxiety disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Effect of wearing a compression vest on patient reported outcome pain | At baseline
  Brief Pain Inventory (BPI) for pain questionnaire
Effect of wearing a compression vest on patient reported outcome pain two weeks after wearing a compression vest | 2 weeks
  Brief Pain Inventory (BPI) for pain questionnaire
Effect of wearing a compression vest on patient reported outcome pain one month after wearing a compression vest | 1 month
  Brief Pain Inventory (BPI) for pain questionnaire
Effect of wearing a compression vest on patient reported outcome pain three months after wearing a compression vest | 3 months
  Brief Pain Inventory (BPI) for pain questionnaire
Effect of wearing a compression vest on patient reported outcome pain six months after wearing a compression vest | 6 months
  Brief Pain Inventory (BPI) for pain questionnaire

SECONDARY OUTCOMES:
Effect of wearing a compression vest on degree of breast edema (CTCAE score) | At baseline
  During each study related visit to the hospital CTCAE score (Common Terminology Criteria for Adverse Events version 4.0) will be registered.
Effect of wearing a compression vest on degree of breast edema (CTCAE score) | At 1 month
  During each study related visit to the hospital CTCAE score (Common Terminology Criteria for Adverse Events version 4.0) will be registered.
Effect of wearing a compression vest on degree of breast edema (CTCAE score) | At 3 months
  During each study related visit to the hospital CTCAE score (Common Terminology Criteria for Adverse Events version 4.0) will be registered.
Effect of wearing a compression vest on degree of breast edema (CTCAE score) | At 6 months
  During each study related visit to the hospital CTCAE score (Common Terminology Criteria for Adverse Events version 4.0) will be registered.
Effect of wearing a compression vest on patient reported quality of life | At baseline
  EORTC QLQ-C30 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 2 weeks after wearing a compression vest
  EORTC QLQ-C30 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 1 month after wearing a compression vest
  EORTC QLQ-C30 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 3 months after wearing a compression vest
  EORTC QLQ-C30 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 6 months after wearing a compression vest
  EORTC QLQ-C30 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At baseline
  EORTC QLQ-BR23 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 2 weeks after wearing a compression vest
  EORTC QLQ-BR23 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 1 month after wearing a compression vest
  EORTC QLQ-BR23 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 3 months after wearing a compression vest
  EORTC QLQ-BR23 for quality of life and breast edema symptoms
Effect of wearing a compression vest on patient reported quality of life | At 6 months after wearing a compression vest
  EORTC QLQ-BR23 for quality of life and breast edema symptoms

IPD SHARING:
Plan to Share IPD: Undecided